CLINICAL TRIAL: NCT04585347
Title: Four-Period, Single-Dose, Sequential Study in Healthy Adults, to Assess Pharmacokinetics of ALZ-801 and Tramiprosate From ALZ-801 Prototype Tablets and Effect of Food on Bioavailability of ALZ-801 and Tramiprosate for Selected Prototype Tablet
Brief Title: Single Dose Study of ALZ-801 Prototype Tablets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Alzheon Inc. (Industry)
Collaborators: Quotient Clinical (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ALZ-801-104
Record Dates: First submitted 2020-10-09; First posted 2020-10-14 (Actual); Last update posted 2020-10-14 (Actual); Status verified 2020-10

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — ALZ-801; Postprandial Period

STUDY DESIGN:
Intervention Model Description: Subjects were to receive a single oral dose of ALZ-801 in each of the 4 study periods (Regimens A, B, C and D) in a non-randomized, sequential manner, separated by a minimum washout period of 7 days.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Regimen A (Experimental): ALZ-801 171 mg tablet, fasting, once
  Interventions: Drug: ALZ-801 170 mg Fasting
- Regimen B (Experimental): ALZ-801 205 mg tablet, fasting, once
  Interventions: Drug: ALZ-801 205 mg Fasting
- Regimen C (Experimental): ALZ-801 205 mg tablet, after food once
  Interventions: Drug: ALZ-801 205 mg After Food
- Regimen D (Experimental): ALZ-801 342 mg (administered as 2 x 171 mg tablets of ALZ-801), after food, once
  Interventions: Drug: ALZ-801 342 mg Fasting

INTERVENTIONS:
Drug: ALZ-801 170 mg Fasting
  Arms: Regimen A
Drug: ALZ-801 205 mg Fasting
  Arms: Regimen B
Drug: ALZ-801 205 mg After Food
  Arms: Regimen C
Drug: ALZ-801 342 mg Fasting
  Arms: Regimen D

SUMMARY:
Phase 1, single-center, open-label, non-randomized, sequential single dose 4-period study in 12 healthy subjects to assess the pharmacokinetics of ALZ-801, tramiprosate and the primary metabolite of tramiprosate, NRM5074, from prototype drug product formulations of ALZ-801, and to assess effect of food on the bioavailability of ALZ-801 and tramiprosate of the prototype tablet formulation.

DETAILED DESCRIPTION:
This is a single-center, open-label, non-randomized, sequential, single-dose, 4-period study in 12 healthy adult subjects. Subjects are to receive a single oral dose of ALZ-801 in each of the 4 study periods (Regimens A, B, C and D) in a non-randomized, sequential manner, separated by a minimum washout period of 7 days. The washout period is expected to last approximately 14 days to permit interim decisions to take place and to allow for the selection of the formulation of the subsequent regimen. Periods of interim analysis will take place following dosing with prototype formulations Regimens A, B, and C, during which the PK and safety data are reviewed to determine the dose to be administered in the subsequent treatment period. Interim decisions aim to identify a prototype ALZ-801 immediate release tablet formulation that provides a similar tramiprosate AUC and Cmax to that of historical values after administration of a 100 mg loose-filled tramiprosate capsule in the fasted state.

Optimization of the required tramiprosate exposure will be made by adjusting the dose of ALZ-801 in the prototype tablets using a formulation design space with a target dose range, per tablet, of 171 to 514 mg ALZ-801 (equivalent to 100 mg to 300 mg tramiprosate). Dose selection will be made after a complete review of all data collected from the previous dose group. For dose selection to occur, data is required to be available from a minimum of 8 evaluable subjects with complete safety assessments up to 24 h post-dose, and required safety and PK data (AEs, plasma concentrations of ALZ-801, tramiprosate and NRM5074, and Tmax, Cmax and AUC estimates for ALZ-801 and tramiprosate).

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and females
* Females must be of non-childbearing potential
* Body mass index (BMI) of 18.0 to 35.0 kg/m2

Exclusion Criteria:

* History of any drug or alcohol abuse in the past 2 years
* Subjects known to have a creatinine clearance of <60 mL/min
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) results
* History of cardiovascular, renal, hepatic, neurological, psychiatric, chronic respiratory or gastrointestinal disease as judged by the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2015-09-16 (Actual); Primary Completion 2015-11-13 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
Cmax for ALZ-801, tramiprosate, and NRM5074 | 72 hours after dosing
  Maximum observed concentration
Tmax for ALZ-801, tramiprosate, and NRM5074 | 72 hours after dosing
  Time from dosing at which Cmax was apparent
AUC for ALZ-801, tramiprosate, and NRM5074 | 72 hours after dosing
  Area under the curve from time zero to the last measurable concentration
T1/2 for ALZ-801, tramiprosate, and NRM5074 | 72 hours after dosing
  The apparent elimination half-lifee
Frel for ALZ-801 and tramiprosate | 72 hours after dosing
  Relative bioavailability of mean PK parameters (AUC[0-inf] and Cmax) for fasted compared to fed state for ALZ-801 and tramiprosate
Frel (test to literature reference) | 72 hours after dosing
  Relative bioavailability of mean PK parameters (AUC[0-inf] and Cmax) for tramiprosate from ALZ-801 prototype tablet formulation compared to previous tramiprosate Phase 3 data

SECONDARY OUTCOMES:
Number of participants with adverse events | 72 hours
  Incidence and nature of adverse events (AEs) and serious adverse events (SAEs). Assessments reported as AEs or SAEs include physical examination, clinical laboratory tests, and 12-lead electrocardiogram (ECG) findings

CONTACTS AND LOCATIONS:
Overall Officials: Ann Church, PhD, Study Director — Quotient Clinical

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hey JA, Yu JY, Versavel M, Abushakra S, Kocis P, Power A, Kaplan PL, Amedio J, Tolar M. Clinical Pharmacokinetics and Safety of ALZ-801, a Novel Prodrug of Tramiprosate in Development for the Treatment of Alzheimer's Disease. Clin Pharmacokinet. 2018 Mar;57(3):315-333. doi: 10.1007/s40262-017-0608-3. PMID 29063518
- See also: Clinical Pharmacokinetics and Safety of ALZ-801 — http://link.springer.com/article/10.1007%2Fs40262-017-0608-3